CLINICAL TRIAL: NCT06808906
Title: The Effect of Hand Massage on Pain, Anxiety, and Comfort Levels of Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva SERT, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAÜ-HAND MASSAGE
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: hand massage; pain; anxiety; comfort; Intensive care unit; nursing
MeSH Terms: conditions — Stroke; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria were divided into two groups: intervention and control. The groups were randomized according to the protocol numbers of the patients in a computerized environment. Patients in the intervention group were informed about the procedure before starting the massage.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Hand massage application steps were based on Kolcaba's Comfort Theory, and the protocol was followed accordingly
  Interventions: Other: Hand Massage Application
- Control (No Intervention): Individuals in the control group did not receive any intervention and received routine nursing care. The patients in the control group were administered VAS, GCS-SF, and STAI twice at 10-minute intervals on the first day after randomization and VAS, GCS-SF, and STAI two weeks later.

INTERVENTIONS:
Other: Hand Massage Application — Hand massage was applied for a total of 12 sessions in two weeks. Care was taken to perform the hand massage application outside the treatment and care hours, and it was performed in a quiet environment. The application was started from the same hand in the same patient in each session, and the same clinic nurse massaged all patients. Since the patients were in the intensive care unit, their vital signs were monitored 24. It was carefully monitored whether there was any change in vital signs during the massage. The patient's hand to be applied was placed on the pillow or bed. Clothes covering the upper extremity starting from the elbow area were removed. The patient was placed in a supine or semi-fowler position. The nurse practitioner took a standing position. She started the massage with effleurage, first on the back of the hand, then on the palm, from the fingertips towards the heart direction, placing the thumbs on the area to be treated and applying effleurage 5 times in a half-mo
  Arms: Intervention

SUMMARY:
This study titled "Evaluation of the Effect of Hand Massage on Patients' Pain, Anxiety and Comfort Levels" aims to determine the effect of hand massage on patients in intensive care units. Our study is single-center and will continue until May 30, 2023. The study is designed to create an experimental and control group. Your patient is in the control group of the study. During the application period of the study, patients in the control group will be provided with routine nursing care and no additional nursing intervention will be applied. Patients in the intervention group of the study will be applied a total of 12 sessions of hand massage, 6 sessions per week (15 minutes each session).

DETAILED DESCRIPTION:
The study sample consisted of patients who were receiving treatment at the Neurology Intensive Care Unit of Sakarya University Training and Research Hospital between April and May 2023, who met the inclusion criteria and agreed to participate in the study. The patients were divided into an intervention group (n=32) that received 15-minute hand massage and a control group (n=32) that received routine nursing care. The Sociodemographic Data Form, Visual Pain Scale (VAS), General Comfort Scale-Short Form and Spielberger State-Trait Anxiety Inventory (STAI) were used to collect data. Inclusion Criteria

* Being 18 years of age or older
* Agreeing to participate in the study and having written permission
* Not having any cognitive, sensory or mental disorders
* Being able to speak and communicate in Turkish
* Being fully oriented to place, time and person
* Individuals to be included should not have conditions such as masses, loss of sensation, fractures or ingrown toenails in their hands

Exclusion Criteria

* Patients who do not agree to participate in the study
* Patients who want to leave the study during the research process will not be included.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and over who agreed to participate in the study
* whose written consent was obtained
* who had no communication problems (hearing, vision, speech, and perception) were included in the study.

Exclusion Criteria:

* Patients who did not agree to participate in the study, who had conditions such as mass in the hand area, sensory loss, previous surgical operation, allergy or skin disease, fracture, and ingrown nail, and who could not complete 12 sessions were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | 15 minutes and 60 minutes after 10 minutes of hand massage
  It is a 10 cm horizontal or vertical line with different numbers on both ends (0=no pain, 10=most severe pain). In many studies, it is used as an easy-to-apply and understandable scale for the assessment of pain intensity. VAS is also used for the assessment of comfort.
General Comfort Scale-Short Form (GCS-SF) | 15 minutes and 60 minutes after 10 minutes of hand massage
  The scale has sub-dimensions of relief (9 items), ease (9 items), and transcendence (10 items). In the evaluation of the scale consisting of positive and negative items, negative items are reverse coded and summed. The highest total score that can be obtained from the scale is 112, and the lowest score is 28
Spielberg State-Trait Anxiety Inventory (STAI) | 15 minutes and 60 minutes after 10 minutes of hand massage
  The scale, which was developed based on the two-factor anxiety concept to determine the state and trait anxiety levels of individuals, consists of a total of 40 items and two separate sections. Two different sections determine transient-state (20 items) and trait (20 items) anxiety levels. The State Anxiety Scale (SAS) determines how the individual feels at a certain moment and in a certain situation, and the Trait Anxiety Scale (TAS) determines how the individual generally feels. A total of 20-80 points are obtained from these scales. The highest score obtained from the scale indicates a high level of anxiety. An increase in the total score obtained from the scale indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No